CLINICAL TRIAL: NCT00942682
Title: Phase I Study of Sorafenib in Combination With RAD001 in Patients With Advanced Neuroendocrine Tumors
Brief Title: Sorafenib in Combination With RAD001 in Patients With Advanced Neuroendocrine Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Novartis (Industry); Bayer (Industry)
Responsible Party: Principal Investigator, Jennifer Chan, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-094
Record Dates: First submitted 2009-07-17; First posted 2009-07-21 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Neuroendocrine Tumor; Carcinoid Tumor; Pancreatic Neuroendocrine Tumor
Keywords: sorafenib; RAD001
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor; Adenoma, Islet Cell | interventions — Sorafenib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib and RAD001 (Experimental): * Since we are looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects in participants that have neuroendocrine tumors, not everyone who participates in this research study will receive the same dose of the study drug. The dose the participant will be given will depend on the number of participants who have been enrolled in the study.
  * Each treatment cycle lasts 28 days. Participants will take RAD001 orally once a day in the morning. Participants will take sorafenib orally twice daily.
  * Participants will remain on this research study as long as they continue to benefit from the study medications.
  Interventions: Drug: Sorafenib; Drug: RAD001

INTERVENTIONS:
Drug: Sorafenib — Taken orally twice daily
Drug: RAD001 — Taken orally once daily in the morning

SUMMARY:
The purpose of this research study is to find out more about the combination of RAD001 and sorafenib such as the safest dose to use, the side effects it may cause, and if the drug is effective for treating neuroendocrine tumors.

DETAILED DESCRIPTION:
* Since we are looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects in participants that have neuroendocrine tumors, not everyone who participates in this research study will receive the same dose of the study drug. The dose the participant will be given will depend on the number of participants who have been enrolled in the study.
* Each treatment cycle lasts 28 days. Participants will take RAD001 orally once a day in the morning. Participants will take sorafenib orally twice daily.
* Initially participants will come to the clinic every other week. At these visits bloodwork will be taken to monitor the participants health. Every 2 months of treatment, participants will have a CT scan or MRI done to see how the medication is working.
* Participants will remain on this research study as long as they continue to benefit from the study medications.

ELIGIBILITY:
Inclusion Criteria:

* Locally unresectable or metastatic neuroendocrine tumor (carcinoid tumor or pancreatic neuroendocrine tumor). Patients must have confirmed low-grade or intermediate-grade neuroendocrine carcinoma. Patients with poorly differentiated neuroendocrine carcinoma, high-grade neuroendocrine carcinoma, adenocarcinoid, goblet cell carcinoid, and small cell carcinoma are not eligible.
* 18 years of age or older
* Minimum of four weeks since any major surgery, completion of radiation, or completion of all prior systemic anticancer therapy. Bevacizumab should not have been received within the prior 6 weeks.
* Prior treatment with chemotherapy is allowed. Patients may not have received prior therapy with RAD001 or sorafenib. There is no limit to the number of prior chemotherapy regimens a patient may have received. Patients may receive concomitant therapy with somatostatin analogs.
* ECOG performance status 0 or 1
* Life expectancy 12 weeks or more
* Adequate bone marrow, liver and renal function as outlined in the protocol
* Fasting serum glycerides and fasting triglycerides as outlined in the protocol
* INR < 1.5 or PT/PTT within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate.
* Women of child bearing potential must have a negative serum pregnancy test within 14 days of the administration of the first study treatment. Women must not be lactating.

Exclusion Criteria:

* Prior treatment with cytotoxic chemotherapy, radiation, immunotherapy, or any investigational drug within the preceding 4 weeks. Bevacizumab should not have been received within the prior 6 weeks.
* Prior treatment with RAD001 or sorafenib
* Patients who have undergone major surgery within 4 weeks prior to study enrollment.
* Chronic treatment with systemic steroids or another immunosuppressive agent
* Patients should not receive immunization with attenuated live vaccines during study period or within 1 week of study entry.
* Known brain metastases
* Patients with prior or concurrent malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, or other adequately treated in situ cancer, or any other cancer from which the patient has been disease free for five years.
* Patients with uncontrolled diabetes mellitis or a fasting plasma glucose > 1.5 ULN
* Patients who have congestive heart failure (NHYA Class III or IV), unstable angina, sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block or a history of acute myocardial infarction within the six months preceding enrollment. No new onset angina within 3 months preceding enrollment. No cardiac ventricular arrhythmia requiring antiarrhythmic therapy.
* Uncontrolled hypertension
* Active clinically serious infection
* Serious non-healing wound, ulcer, or bone fracture
* Evidence of history of bleeding diathesis or coagulopathy
* Patients with the presence of active or suspected acute or chronic uncontrolled infection or with a history of immunocompromise, including a positive HIV test result
* Patients who have any severe and/or uncontrolled medical conditions or other conditions what could affect their participation in the study
* Use of St. John's Wort or rifampin (rifampicin)
* Patients with a known or suspected hypersensitivity to sorafenib, RAD001 or other rapamycins or to its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) for sorafenib in combination with RAD001 in patients with advanced neuroendocrine tumors. | 2 years
To determine the dose-limiting toxicities of sorafenib combined with RAD001 in patients with advanced neuroendocrine tumors | 2 years

SECONDARY OUTCOMES:
To determine the safety and tolerability of the combination of sorafenib and RAD001 in patients with advanced neuroendocrine tumors. | 2 years
To make a preliminary assessment of the anti-tumor activity of the combination of sorafenib and RAD001 in patients with advanced neuroendocrine tumors. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Chan, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Result] Chan JA, Mayer RJ, Jackson N, Malinowski P, Regan E, Kulke MH. Phase I study of sorafenib in combination with everolimus (RAD001) in patients with advanced neuroendocrine tumors. Cancer Chemother Pharmacol. 2013 May;71(5):1241-6. doi: 10.1007/s00280-013-2118-9. Epub 2013 Mar 9. PMID 23475104